CLINICAL TRIAL: NCT07354139
Title: Examining Speech Production Errors in Stuttering Through High Definition - Transcranial Direct Current Stimulation
Brief Title: Using Non-invasive Brain Stimulation to Explore Potential Treatments to Reduce Speech Errors in Adults Who Stutter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Principal Investigator, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-25-184
Record Dates: First submitted 2026-01-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stuttering; Fluency Disorder
Keywords: Stuttering; HD-tDCS; neuromodulation; speech; fluency
MeSH Terms: conditions — Stuttering; Speech | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Left Inferior Frontal Gyrus (Experimental): This arm is designed to analyze if treatment on the speech production area of the brain (also known as Broca's area) will decrease speech errors and increase ease of production in people who stutter
  Interventions: Device: High - Definition Transcranial Direct Current Stimulation
- Presupplementary motor area (Experimental): This arm is designed to investigate whether treatment targeting the motor planning region of the brain can reduce speech errors and increase ease of production in individuals who stutter.
  Interventions: Device: High - Definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High - Definition Transcranial Direct Current Stimulation — HD-tDCS protocol for LIFG group is as follows: A single 20-minute session with one anode at F7 at 1 mA and four 0.25 mA cathodes at T7, FP1, AF3, FC5 at 0.25 mA
  HD-tDCS protocol for the Pre-SMA group is as follows: A single 20-minute session with one anode 1mA at Fz 1 mA and four 0.25 mA cathodes at FP1, FP2, F7, F8
  Other Names: Neuroelectrics; Starstim; HD-tDCS; Non-invasive brain stimulation; neuromodulation

SUMMARY:
The goal of this study is to find out whether a type of noninvasive brain stimulation can help reduce speech errors, such as repetitions, blocks, and prolongations, in people who stutter. This pilot study will help researchers design future treatments to see if targeting certain brain areas can improve speech fluency. The study will look at how people speak and behave during both speaking and non-speaking tasks before and after the brain stimulation.

Participants will complete an online survey about 24 hours before coming to the clinic. The clinic visit will last about 3 hours and will include three phases. All parts of the study will be audio-recorded.

1. Pre-Testing: Participants will first complete a stuttering evaluation to determine whether they are typical speakers or have a mild, moderate, or severe stutter. Then, they will do several speaking and non-speaking tasks.
2. Brain Stimulation: Participants will receive a session of targeted noninvasive brain stimulation (HD-tDCS).
3. Post-Testing: After the brain stimulation, participants will repeat the same evaluation and tasks they completed during pre-testing.

Brain stimulation description:

HD-tDCS is a non-invasive technique that requires the placement of several sensors (metal electrodes) on a special cap and saline gel on your head. Very low levels of constant electrical current are delivered to specifically targeted areas of the brain via these electrodes. You may experience a slight feeling of dizziness when starting the stimulation. This occurs in a small number of subjects. This takes only a few seconds and does not affect balance after the stimulation has been completed. Several research centers have previously investigated the use of this device on healthy subjects and have found the device to be safe with no direct effect on the person's well-being. Following stimulation, participants will have the opportunity to rinse out residual gel from hair and scalp.

ELIGIBILITY:
Inclusion Criteria:

* Must be 22 years old or older
* May be bi/multilingual but must speak English as dominant language.
* Must be diagnosed or suspected of developmental stuttering disorder. Participants will be administered the Stuttering Severity Instrument 4 and categorized as typical speakers or mild, moderate, or severe stutterers.
* Must be able to attend the session at the physical location within the clinic

Exclusion Criteria:

* Patients with preexisting speech/language disorders or previously diagnosed neurological disorders (including but not limited to apraxia of speech, cerebral palsy, dysarthria, tourettes, or any other neurological/motor condition) that affect speech/language (except stuttering) are excluded to minimize the interference of atypical brain activity.
* Participants who have acquired or neurogenic stuttering (stuttering resulting from a brain injury) are excluded, as this study focuses exclusively on the effects of developmental stuttering.
* Participants with a history of seizures
* Participants with unexplained episodes of loss of consciousness, since such condition could be related with brain alterations or epilepsy
* Participants with unstable or non controlled neuropsychiatric illness
* Participants having implanted brain medical devices
* Participants with implanted pacemakers
* Participants having any electrically,magnetically or mechanically activated implant
* Participants having cardiac, neural or medication implants
* Participants having vascular clips or any other electrically sensitive support system in the brain
* Participants with serious brain injury
* Participants showing damage of skin at sites of stimulation (the device can only be used in healthy skin without wounds, otherwise the resistance to current can be altered)
* Participants suffering from skin problems, such as dermatitis, psoriasis or eczema
* Participants suffering from severe or frequent headaches
* Participants with any serious life-threatening disease such as congestive heart failure, pulmonary obstructive chronic disease, or active neoplasia
* Pregnant women
* Participants may not consume alcohol or controlled substances within 24 hours of the scheduled appointment

Participants will complete an additional screener upon enrollment to assess medical history and current drug/medication use that may conflict with the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Stuttering Severity Instrument - 4 | Measured at singular clinical visit (baseline)
  Stuttering Severity Instrument-Fourth Edition (SSI-4) is a reliable and valid norm-referenced stuttering assessment that can be used for both clinical and research purposes. It measures stuttering severity in both children and adults in the four areas of speech behavior:
  frequency duration physical concomitants naturalness of the individual's speech.
  The SSI-4 scores stuttering severity by combining measures of frequency (% syllables stuttered), duration (length of longest stutters), and physical concomitants (secondary behaviors) into a total score, which is then converted to a percentile rank and severity level (very mild to very severe) using age-specific standards. Higher percentile scores indicate more severe stuttering, with ranges like 1-4% being very mild and 96-99% very severe.
Predictive Naming Task | Measured at singular clinical visit (baseline)
  Participants are instructed to name images on a screen, given phrases that indicate high or low predictability for the target word.
  Task is measured by accuracy (number of correct answers) and participant response time.

SECONDARY OUTCOMES:
Overall Assessment of the Speaker's Experience of Stuttering | Completed during enrollment process (24 hours pre-visit during consent)
  The Overall Assessment of the Speaker's Experience of Stuttering (OASES) gives clinicians and researchers an impact rating and impact score, which reflect the degree of adverse impact a speaker experiences due to stuttering. The impact score combines information about (a) the speaker's perceptions about stuttering; (b) the negative affective (feelings), behavioral (actions), and cognitive (thoughts) reactions that the speaker has to stuttering; (c) the functional communication difficulties a speaker may have in different speaking environments; and (d) the impact of stuttering on the speaker's overall quality of life. The OASES is the only published tool that specifically examines Quality of Life in people who stutter.
  The OASES score reflects the impact of stuttering on a person's life, using a 1-5 rating scale where higher scores indicate a more severe impact, categorized into mild, mild-to-moderate, moderate, moderate-to-severe, and severe levels.
Button push Go/NoGo task | Measured at singular clinical visit (baseline)
  Participants are instructed to press a button when category A (objects) is presented on the screen, but not to push when category B (animals) is shown.
  Task is measured by accuracy (number of correct answers) and participant response time.

CONTACTS AND LOCATIONS:
Locations (1):
- Callier Clinical Research Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and clinical study report will be available for the public
Supporting Information: CSR
Time Frame: IPD data will be available 3 months after publication
Access Criteria: The Clinical Study Report (CSR) will be made available upon reasonable request. Researchers must submit a brief written request describing the purpose of accessing the CSR. Requests will be reviewed by the study team for appropriateness and compliance with institutional policies.